CLINICAL TRIAL: NCT05454969
Title: Transforming Healthcare in Post-Pandemic Recovery: Innovation in Process & Technology to Increase Patient Throughput While Reducing Clinician Burden and Addressing Health Disparities (One-4-ALL Initiative)
Brief Title: One-4-ALL Initiative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0995
Record Dates: First submitted 2022-06-27; First posted 2022-07-12 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Literacy; Burden, Caregiver; Health Care Utilization
MeSH Terms: conditions — Literacy; Caregiver Burden; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial to examine pre-post differences between individuals that use the app versus the standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-4-ALL Initiative (Active Comparator): The health app arm will pilot the intervention and key outcome measures will be compared between the Health App group and the placebo control.
  Interventions: Behavioral: One-4-ALL Initiative
- Control (Placebo Comparator): Will receive standard care.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: One-4-ALL Initiative — We can successfully implement a patient app that will be used by families to 1) increase throughput for all patients, including minoritized, low-income, and low health literacy patients, and 2) reduce administrative burdens on providers.
  Arms: One-4-ALL Initiative
Behavioral: Control — Patients will receive standard of care.
  Arms: Control

SUMMARY:
This study aims to improve health outcomes of individuals and populations, enhance the patient experience, reduce the per capita cost of care, and ensure the well-being of our healthcare providers (quadruple aim). These goals are increasingly difficult to achieve, given the challenges of changes to workflow, staffing shortages, and increased costs brought on by the COVID-19 pandemic. Further, the pandemic brought to light the critical need to transform healthcare access for our racially and culturally minoritized and low-income families that have long been victims of health disparities, specifically with poorer health outcomes.

DETAILED DESCRIPTION:
The overall objective is to successfully implement a patient app that will be used by families to 1) increase throughput for all patients, including minoritized, low-income, and low health literacy patients, and 2) reduce administrative burdens on providers.

To evaluate this hypothesis, the following specific aims will be examined:

Aim 1: Document modifiable factors that negatively and positively impact providers' ability to provide high-quality patient care in a post-pandemic healthcare system while addressing health disparities through implementation science.

Aim 2: Create a "boarding pass' experience for providers and patients using technology (app) which allows patients and their families to fully prepare for their clinical visits and bridge care between home, primary care providers, and specialty care.

Aim 3: Investigate multilevel contextual factors related to app implementation, to inform future strategies to promote scalability and sustainability of app in all specialties.

ELIGIBILITY:
Inclusion Criteria:

* All guardians of patients and the providers (surgeons, doctors, nurses, etc) that serve these patients.

Exclusion Criteria:

* None.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Health care quality | post-intervention (12 weeks)
  Health care quality will be assessed using six domains; safety, effective, patient-centered, timely, efficient, and equitable. Likert scale 1-5, higher score is best.
Provider satisfaction | post-intervention (12 weeks)
  Provider job satisfaction including level of burden and overall job satisfaction. Likert scale 1-5, higher score is best.
  physical and mental health
Patient satisfaction | post-intervention (12 weeks)
  Patient's satisfaction of the program tool. Likert scale 1-5, higher score is best.
  literacy of the patient & their family, patient & family anxiety pre-surgery.
Acceptability of program tool | post-intervention (12 weeks)
  Patient's ability to engage and understand the program tool. Likert scale 1-5, higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Landsbaugh Kaar, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No